CLINICAL TRIAL: NCT01557699
Title: An Open-Label, Randomized, Phase I Study in Healthy Male Adults to Evaluate the Safety of a Measles Vaccine (Dry Powder)Administered by Two Devices
Brief Title: A Clinical Trial to Assess the Safety of a Measles Vaccine (Dry Powder) Administered by Two Different Devices
Acronym: PMV-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: University of Colorado, Boulder (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PMV-001; CTRI/2012/02/002447 (Registry Identifier: CLINICAL TRIAL REGISTRY OF INDIA (CTRI))
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Prophylaxis for the Measles Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PMV via Puffhaler® Device (Experimental): The dry powder measles vaccine will be administered via a Puffhaler® device. A single dose of 10 mg will be used.
  Interventions: Biological: PMV via Puffhaler® device
- PMV via SoloventTM device (Experimental): The dry powder measles vaccine will be administered via a SoloventTM device. A single dose of 10 mg will be used.
  Interventions: Biological: PMV via SoloventTM device
- Licensed Subcutaneous Measles Vaccine (Active Comparator): Licensed measles vaccine will be administered subcutaneously as single dose of 0.5 ml.
  Interventions: Biological: Licensed Subcutaneous Measles Vaccine

INTERVENTIONS:
Biological: PMV via Puffhaler® device — The vaccine will be administered via a Puffhaler® device. A single dose of 10 mg of PMV (dry powder measles vaccine) will be used.
  Arms: PMV via Puffhaler® Device
Biological: PMV via SoloventTM device — The vaccine will be administered via SoloventTM device. A single dose of 10 mg of PMV (dry powder measles vaccine) will be used.
  Arms: PMV via SoloventTM device
Biological: Licensed Subcutaneous Measles Vaccine — This is a licensed formulation containing the live attenuated Edmonston Zagreb virus. A single dose of 0.5 ml will be given subcutaneously.
  Other Names: SMV
  Arms: Licensed Subcutaneous Measles Vaccine

SUMMARY:
This is a phase I, open-label, randomized study in healthy adults. Eligible subjects will be given single dose of either Dry Powdered Measles Vaccine (PMV) by Puffhaler® device, Dry PMV by SoloventTM device or licensed measles vaccine by subcutaneous route (SMV). Subjects will be followed for 180 days for safety.

DETAILED DESCRIPTION:
This is a phase I, open-label, randomized study in healthy adults. Eligible subjects will be given single dose of either Dry Powdered Measles Vaccine (PMV) by Puffhaler® device, Dry PMV by SoloventTM device or licensed measles vaccine by subcutaneous route (SMV). Solicited reactions will be assessed for first 14 days after vaccination and unsolicited adverse events will be assessed till 84 days after vaccination. Subjects will be followed for 180 days for any SAEs.

ELIGIBILITY:
Inclusion Criteria:

* Male adults of age of 18-45 years.
* Measles immune, as determined by IgG antibody levels.
* Healthy as supported by medical history, physical examination and laboratory evaluation on preset parameters.
* Signed informed consent for participation in trial and for HIV screening.

Exclusion Criteria:

* Medical history of immunodeficiency/suppression or subject with history of close contact with immunocompromised/ immunosuppressed person.
* Chronic administration of immunosuppressants or other immune modifying agents
* Acute febrile illness or suspected measles illness or acute infectious disease
* Acute or chronic, clinically significant pulmonary, endocrine, autoimmune, psychiatric, cardiovascular, neurological, hepatic or renal functional abnormality which in the opinion of the investigator, might interfere with the study objectives
* History of seizure disorders
* Major congenital defects
* Thrombocytopenia or known bleeding disorders 8. History of a previous severe allergic reaction
* Positive serology for HIV antibody, HCV antibody or Hepatitis B surface antigen
* Known hypersensitivity to any component of the study vaccine

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharad Agarkhedkar, MD, Principal Investigator — Department of Pediatrics, Padmashree Dr. D. Y. Patil Medical College Hospital & Research Centre, Sant Tukaram Nagar, Pimpri Pune-411018
Locations (1):
- Department of Pediatrics, Padmashree Dr. D. Y. Patil Medical College, Pune, Maharashtra, India

REFERENCES:
- [Result] MVDP author group; Cape S, Chaudhari A, Vaidya V, Mulay R, Agarkhedkar S, Shermer C, Collins M, Anderson R, Agarkhedkar S, Kulkarni PS, Winston S, Sievers R, Dhere RM, Gunale B, Powell K, Rota PA, Papania M. Safety and immunogenicity of dry powder measles vaccine administered by inhalation: a randomized controlled Phase I clinical trial. Vaccine. 2014 Nov 28;32(50):6791-7. doi: 10.1016/j.vaccine.2014.09.071. Epub 2014 Oct 22. PMID 25446830

RESULTS

PARTICIPANT FLOW:
Groups:
- Dry Powdered Measles Vaccine Via a Puffhaler® Device: Dry Powdered Measles Vaccine: The vaccine was administered via a Puffhaler® device. A single dose of 10 mg was used.
  N=20
- Dry Powdered Measles Vaccine Via SoloventTM Device: Dry Powdered Measles Vaccine: The vaccine was administered via SoloventTM device. A single dose of 10 mg was used.
  N=20
- Licensed Subcutaneous Measles Vaccine: Licensed Subcutaneous Measles Vaccine: This is a licensed formulation containing the live attenuated Edmonston Zagreb virus. A single dose of 0.5 ml was given subcutaneously.
  N=20
Period: Overall Study
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 60 healthy adult males of 18 to 45 years
Groups:
- PMV Puffhaler®: Dry Powdered Measles Vaccine: The vaccine was administered via a Puffhaler® device. A single dose of 10 mg was used.
  N=20
- PMV SoloventTM: Dry Powdered Measles Vaccine: The vaccine was administered via SoloventTM device. A single dose of 10 mg was used.
  N=20
- Subcutaneous Meales Vaccine: Licensed Subcutaneous Measles Vaccine: This is a licensed formulation containing the live attenuated Edmonston Zagreb virus. A single dose of 0.5 ml was given subcutaneously.
  N=20
- Total: Total of all reporting groups
Arm/Group | PMV Puffhaler® | PMV SoloventTM | Subcutaneous Meales Vaccine | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7) [18 to 45] | 30 (6) | 28 (7) | 28.67 (6.67)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: Male participants] | 20 | 20 | 20 | 60
Region of Enrollment [Number; unit: participants]
  India | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Solicited Reactions
Description: Incidence of solicited local and systemic reactions within 14 days of vaccine administration in each group was assessed.
Time Frame: Day 14
Population: Intention-To-Treat (ITT) Population included all subjects who received at least one dose of study vaccine and had at least one post-baseline assessment, regardless of whether they adhered to the study eligibility criteria or whether their study medication administration and study procedure visits are within the protocol-specified windows.
Measure: Number; unit: participants
Groups:
- PMV Puffhaler®: Dry Powdered Measles Vaccine: The vaccine was administered via a Puffhaler® device. A single dose of 10 mg was used.
- PMV SoloventTM: Dry Powdered Measles Vaccine: The vaccine was administered via SoloventTM device. A single dose of 10 mg was used.
- Subcutaneous Meales Vaccine: Licensed Subcutaneous Measles Vaccine was administered as single dose of 0.5 ml subcutaneously
Arm/Group | PMV Puffhaler® | PMV SoloventTM | Subcutaneous Meales Vaccine
Number analyzed (Participants) | 20 | 20 | 20
participants | 0 | 0 | 0

2. Primary Outcome: Incidence of Unsolicited Adverse Events Within 84 Days
Description: Incidence of unsolicited adverse events for a period of 84 days in each group was assessed.
Time Frame: Day 84
Population: Intention-To-Treat (ITT) Population was used for safety analysis.
Measure: Number; unit: participants
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Number analyzed (Participants) | 20 | 20 | 20
participants | 0 | 0 | 0

3. Primary Outcome: Incidence of Serious Adverse Events (SAEs) and New Onset Chronic Medical Conditions
Description: Incidence of serious adverse events (SAEs) and new onset chronic medical conditions throughout the entire study period of 180 days in each group was assessed.
Time Frame: Day 180
Population: Intention-To-Treat (ITT) Population was used for safety and immunogenicity analysis. ITT population included subjects who had blood drawn to confirm a measles protective titer at Day -7 and met all inclusion/ exclusion criteria and did not receive a vaccine forbidden in the study protocol within the previous 30 days.
Measure: Number; unit: participants
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Number analyzed (Participants) | 20 | 20 | 20
participants | 0 | 0 | 0

4. Secondary Outcome: The Proportion of Subjects in Each Group With Seropositive Anti-Measles IgG Antibodies
Description: The proportion of subjects in each group with seropositive anti-Measles IgG antibodies on Day -7, Day 28 and Day 84 was assessed.
Time Frame: Day -7, Day 28 and Day 84
Population: Per Protocol (PP) Population was for the Immunogenicity analysis & included subjects who received a dose of the study vaccine and met all inclusion/ exclusion criteria and complied with study procedures as defined in the study protocol, did not show any major protocol violation and gave baseline (Day -7) and Day 28 immunogenicity blood samples.
Measure: Number; unit: percentage of participants
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Number analyzed (Participants) | 20 | 20 | 20
percentage of participants | 100 | 100 | 100

5. Secondary Outcome: The Proportion of Subjects in Each Group With Seroprotective Plaque-reduction Neutralization Test (PRNT) Titre
Description: The proportion of subjects in each group with seroprotective plaque-reduction neutralization test (PRNT) titre on Day -7, Day 28 and Day 84 was assessed.
Time Frame: Day -7, Day 28 and Day 84
Population: Per Protocol (PP) Population was used for the Immunogenicity analysis which included subjects who received a dose of the study vaccine and met all inclusion/ exclusion criteria and complied with study procedures as defined in the study protocol, did not show any major protocol violation and gave baseline (Day -7) and Day 28 blood samples.
Measure: Number; unit: percentage of participants
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Number analyzed (Participants) | 20 | 20 | 20
percentage of participants | 100 | 100 | 95

6. Secondary Outcome: The Proportion of Subjects in Each Group With Seroconversion for Serum Anti-Measles IgG
Description: The proportion of subjects in each group who show a seroconversion for serum anti-Measles IgG on Day 28 and Day 84 was assessed.
Time Frame: Day 28 and Day 84
Population: Per Protocol Population was used for the Immunogenicity analysis which included subjects who received a dose of the study vaccine and met all inclusion/ exclusion criteria and complied with study procedures as defined in the study protocol, did not show any major protocol violation and gave baseline (Day -7) and Day 28 blood samples.
Measure: Number; unit: percentage of participants
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Number analyzed (Participants) | 20 | 20 | 20
percentage of participants
  at day 28 | 45 | 20 | 25
  at day 84 | 55 | 45 | 35

7. Secondary Outcome: The Proportion of Subjects in Each Group With Seroconversion for PRNT
Description: The proportion of subjects in each group who show a seroconversion for PRNT on Day 28 and Day 84 was assessed.
Time Frame: Day 28 and Day 84
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Number analyzed (Participants) | 20 | 20 | 20
percentage of participants
  Day 28 | 45 | 25 | 30
  Day 84 | 30 | 30 | 25

8. Secondary Outcome: Geometric Mean Concentration (GMC) for Anti-Measles IgG Antibodies
Description: Geometric Mean Concentration (GMC) for anti-Measles IgG antibodies were measured on Day -7, Day 28 and Day 84 by ELISA using Trinity ELISA Kits for Measles.
Time Frame: Day -7, Day 28 and Day 84
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Number analyzed (Participants) | 20 | 20 | 20
IU/ml
  Baseline (Day-7) | 0.91 [0.63 to 1.33] | 1.31 [0.93 to 1.84] | 0.86 [0.57 to 1.32]
  Day 28 | 1.46 [1.06 to 2.01] | 1.49 [1.13 to 1.96] | 1.03 [0.86 to 1.23]
  Day 84 | 1.71 [1.31 to 2.22] | 2.14 [1.72 to 2.68] | 1.45 [1.07 to 1.95]

9. Secondary Outcome: Geometric Mean Titre (GMT) by PRNT on Day -7, 28 and 84
Description: Geometric Mean Titre by Plaque Reduction Neutralization Test were assessed on Day -7, 28 and 84 at CDC, Atlanta. Titers are expressed as IU/ml.
Time Frame: Day -7, Day 28 and Day 84
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Number analyzed (Participants) | 20 | 20 | 20
IU/ml
  Baseline (Day -7) | 1914.3 [826.95 to 4431.6] | 1479.5 [768.41 to 2848.6] | 2010.4 [1033.6 to 3910.5]
  Day 28 | 2626.5 [1719.7 to 4011.4] | 1569.1 [937.44 to 2626.4] | 1789.7 [1047.8 to 3057.0]
  Day 84 | 1789.5 [966.32 to 3313.9] | 1526.5 [824.95 to 2824.8] | 1152.2 [669.71 to 1982.2]

ADVERSE EVENTS:
Time Frame: Day 84
Description: Occurrence of unsolicited adverse events was monitored till day 84 after randomization. No unsolicited adverse events were reported. Subjects had study site visits till day 84. Day 180 visit was telephonic communication with the study subjects to assess if any serious adverse events occurred from day 84 till day 180 after randomization.
Groups:
- Dry Powdered Measles Vaccine Via a Puffhaler® Device: Dry Powdered Measles Vaccine: The vaccine will be administered via a Puffhaler® device. A single dose of 10 mg will be used.
  N=20
- Dry Powdered Measles Vaccine Via SoloventTM Device: Dry Powdered Measles Vaccine: The vaccine will be administered via SoloventTM device. A single dose of 10 mg will be used.
  N=20
- Licensed Subcutaneous Measles Vaccine: Licensed Subcutaneous Measles Vaccine: This is a licensed formulation containing the live attenuated Edmonston Zagreb virus. A single dose of 0.5 ml will be given subcutaneously.
  N=20
Arm/Group | Dry Powdered Measles Vaccine Via a Puffhaler® Device | Dry Powdered Measles Vaccine Via SoloventTM Device | Licensed Subcutaneous Measles Vaccine
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No